CLINICAL TRIAL: NCT06714929
Title: Advancing Water Security: A Community Participatory School-Based Hydration Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: HM20028646; R01HD114792 (NIH)
Record Dates: First submitted 2024-11-10; First posted 2024-12-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Dental Caries; Obesity Prevention
Keywords: hydration; water; sugar-sweetened beverages; dental caries; overweight and obesity
MeSH Terms: conditions — Dental Caries; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized controlled trial; 4 groups of schools sequentially receive the intervention each year over 3 years. Assessments of all 12 schools occur at all timepoints over the 3 years.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Assessment only
- Hydration Intervention (Experimental): 4-month community participatory school-based hydration intervention that includes provision of refillable water bottles in schools with hydration stations in addition to: 1) social marketing, 2) behavioral reinforcement, and 3) education and outreach.
  Interventions: Behavioral: Hydration

INTERVENTIONS:
Behavioral: Hydration — Clusters of schools will sequentially be exposed to the intervention in a stepped-wedge fashion. The intervention is a 4-month community participatory school-based hydration intervention that includes provision of refillable water bottles in schools with hydration stations in addition to: 1) social marketing, 2) behavioral reinforcement, and 3) education and outreach.
  Arms: Hydration Intervention

SUMMARY:
The goal of this study is to determine the effectiveness and sustainability of a community-participatory hydration intervention over 3 years within a district that has newly installed hydration stations and is operating under a policy designed to enhance heathy hydration practices and promote equitable access to drinking water.

DETAILED DESCRIPTION:
The goal of this study is to determine the effectiveness of a hydration intervention on hydration station usage (primary outcome), Body Mass Index z-scores (zBMI) and dental caries (primary biomedical outcomes), and water bottle usage, beverage selection and intake, and academic outcomes (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Lunchroom observations: All students (K-5th [Pre-Kindergarten if applicable]) who eat lunch in the cafeteria on assessment days are eligible
* BMI and dental caries assessments: 1) student enrolls in study while in 3rd grade (followed through 5th g)
* Student surveys: Students in 4th-5th grade are eligible to complete surveys assessing beverage intake and perceptions of hydration practices within their school district.
* Staff surveys: All staff in the target schools will be eligible to complete the Personnel Survey.

Exclusion Criteria:

* Lunchroom observations: None.
* BMI and dental caries assessments: Students are ineligible if they are unable to complete assessments due to developmental or physical reasons, 2) planning to move in the study duration
* Student surveys: None.
* Staff surveys: None.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Water Station Usage | Years 1-3
  Ounces of water per student per day measured by hydration station flow meters.
Dental Caries Status | up to 3 years
  Tooth decay or cavities will be measured using a modified International Caries Detection and Assessment System (ICDAS)
Body Mass Index (BMI) | up to 3 years
  NHANES Anthropometry methods used to measure height and weight. Age and sex-specific BMIz-score and BMI percentile will be calculated using Epi Info

SECONDARY OUTCOMES:
Water Bottle Usage at Lunch | up to 3 years
  % of students with water bottles in school
Beverage Selection at Lunch | up to 3 years
  % of each beverage selected (water, white milk, flavored milk, 100% juice, soda, sports-drink, other sugar-sweetened beverage (SSB), other non-SSB, unknown)
Academics | up to 3 years
  Standards of Learning scores ranging from 0-600 with higher scores representing higher academic proficiency.
Beverage Intake | up to 3 years
  modified beverage intake questionnaire (BEVQ; 12-item) will assess frequency and amount of SSB and water consumption to determine average daily consumption in fl oz and kcal over the past month for each item and across categories: water, total SSBs (sweetened juice and drinks, regular carbonated beverages, sweet tea, sweetened coffee, energy drinks), milk, 100% juice.
Water Source Assessment | up to 3 years
  Video of water sources and then coded by trained raters. Coding for: cleanliness, wear, availability of drinking vessels, filter status, obstructions, signage, trash, and water flow
School Personnel Knowledge | up to 3 years
  Measured via surveys: perceptions of water bottle use and hydration in school, knowledge and beliefs about hydration, personnel hydration practices, and awareness of and adherence to existing hydration policy
School Environment | up to 3 years
  Measured via semi-structured interview: assessing water and SSB-related access, policies and practices in their school
Beverage Sales | up to 3 years
  We will evaluate purchases of white milk, sugar-sweetened milk, 100% juice, and other beverages.
National School Lunch Program (NSLP) Participation | up to 3 years
  Daily and monthly NSLP participation rates will be obtained

OTHER OUTCOMES:
Demographics | up to 3 years
  School-level sex, race, ethnicity and enrollment will be obtained from the Department of Education
Attendance | Pre-intervention, Month 1, Month 2, Month 3
  Attendance by grade on observation days will be obtained (to determine participation rates)
Implementation of Intervention | through study completion, an average of each year
  Fidelity checklists, surveys, logs of implementation components
Perspectives of the intervention | 4 months and 16 months post-intervention
  Semi-structured interviews with key stakeholders to assess barriers and facilitators to intervention implementation and sustainability.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The following research data will be generated from this study: 1) lunchroom observations (beverage selection and water bottle use); 2) cafeteria sales data; 3) hydration station usage; 4) academic data (Standards of Learning scores, attendance); and 4) survey data. Student survey data include demographics, beverage intake, and intervention perceptions. Staff survey data includes hydration policies and practices and intervention perceptions. Longitudinal assessments of anthropometrics (serial height and weight measurements) and dental caries will be available from a subset of students (n=406). A subset of individuals will also complete interviews (n=80) regarding intervention implementation and sustainability. Any potentially identifying information (e.g., of individuals, schools, or the district) will be removed from these data prior to uploading them to the NICHD Data and Specimen Hub.
Supporting Information: Study Protocol, ICF
Time Frame: Final submission and release of the study data will occur no later than the time of an associated publication or end of the performance period, whichever comes first. Study data deposited in DASH are available to the research community in perpetuity.
Access Criteria: Public Use Data: All deidentified study data will be made available as public use data to the research community via DASH. Sharing will occur in accordance with the participant consent and Virginia Commonwealth University (VCU) Institutional Review Board approval. Users of the public use data must register with DASH and agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads. Datasets in DASH will be findable and identifiable through a study digital object identifier (DOI) assigned by DASH.